CLINICAL TRIAL: NCT05672407
Title: The Role of Local Tranexamic Acid on Periorbital Oculoplastic Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Research team dissembled because of no funding.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wendy Lee, Professor of Clinical Ophthalmology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20220736
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Eyelid Diseases; Periorbital Disorder; Hemorrhage; Surgical Blood Loss
MeSH Terms: conditions — Eyelid Diseases; Hemorrhage; Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid Group (Experimental): Participants undergoing standard of care periorbital procedures will be randomized to receive tranexamic acid with lidocaine/epinephrine on one of their eyelids at the beginning of the scheduled operation before incision.
  Interventions: Drug: Tranexamic acid
- Placebo Group (Placebo Comparator): Participants undergoing standard of care periorbital procedures will be randomized to receive balanced salt solution with lidocaine/epinephrine on one of their eyelids at the beginning of the scheduled operation before incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — 100 mg/mL Tranexamic acid with lidocaine with 1:100,000 epinephrine in 1:1 manner administered subcutaneously
  Arms: Tranexamic Acid Group
Drug: Placebo — Lidocaine with 1:100,000 epinephrine mixed with 1:1 Basal Saline Solution (BSS) administered subcutaneously
  Other Names: Balanced Saline Solution
  Arms: Placebo Group

SUMMARY:
This study investigates the effect of tranexamic acid, a medication that helps reduce bleeding, in patients undergoing surgeries around their eyes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above undergoing periorbital oculoplastic surgery including but not limited to upper and lower blepharoplasty, four lid procedures, or dacryocystorhinostomy (DCR).

Exclusion Criteria:

* - Adults unable to consent
* Individuals less than 18 years of age
* Prisoners
* Pregnant women.
* Known contradictions or sensitivities to study medication (tranexamic acid)
* Patients with known prior thromboembolic events
* Previous eyelid surgery or same-side DCR (RE-DCR)
* Has any type of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative patient ecchymosis | Up to 3 months
  Ecchymosis will be graded 0-3 based on location and degree based on a previously reported validated scale (higher scores with more ecchymosis)

SECONDARY OUTCOMES:
Postoperative patient chemosis | Up to 3 months
  Chemosis, swelling of the eyes, will be measured on a scale of 0-4 (higher scores, more edema)
Eyelid edema | Up to 3 months
  Measurement includes through Surgeon Periorbital Ration of Edema and Ecchymosis (SPREE), which has a total score ranging from 1 to 4 with the higher score indicating more severe eyelid edema.
Intraoperative patient bleeding | Postoperative day 0 (day of surgery)
  The amount of blood loss intraoperatively will be measured using a scale for blood soaked materials.
Physician Perception of Intraoperative Bleeding | Postoperative day 0 (day of surgery)
  The primary surgeon will subjectively rank the efficacy of hemostasis on a scale of 1-4 [excellent (1), good (2), moderate (3), or poor (4) ] immediately after the operation.
Patient-perceived outcomes | Up to 3 months
  Patients will complete a validated FACE-Q survey which has a raw score converted to a scaled score of from 0-100, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy W Lee, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No